CLINICAL TRIAL: NCT05393843
Title: Prevention of Maternal and Fetal Metabolic Complications With Polyphenols and Omega-3 Fatty Acids Supplementation in Pregnant Women Affected by Gestational Diabetes on Diet Therapy: a Randomized, Double-blind Placebo Controlled Trial.
Brief Title: Prevention of Maternal and Fetal Metabolic Complications With Diet and Nutraceutical Supplementation in Pregnant Women Affected by Gestational Diabetes: a Randomized, Double-blind Placebo Controlled Trial.
Acronym: PREDIP2
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: outbreak of covid pandemic that caused problems with nutritional coaching in person.
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRE.D.I.P.2
Record Dates: First submitted 2022-05-18; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2018-03

CONDITIONS: Gestational Diabetes; Oxidative Stress
MeSH Terms: conditions — Diabetes, Gestational | interventions — Fatty Acids, Omega-3; Anthocyanins; alpha-Cyclodextrins; Diet

STUDY DESIGN:
Intervention Model Description: randomized, double-blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Active Comparator): patients receiving
  * diet
  * Omega-3 fatty acids (EnerZona Omega3Rx®, Enervit, Italia), at a daily dosage of 2.4 gr at breakfast.
  * Anthocyanins (EnerZona Maqui Response Buste®, Enervit, Italia) at a total daily dosage of 108 mg divided into three equal intakes at breakfast, lunch and dinner.
  * Alpha-cyclodextrins (EnerZona Maqui Response Buste®, Enervit, Italia) at a total daily dosage of 15 gr divided into three equal intakes at breakfast, lunch and din-ner
  Interventions: Dietary Supplement: omega-3 fatty acids, anthocyanins and alpha-cyclodextrins; Behavioral: diet
- placebo (Placebo Comparator): patients receiving
  * diet
  * placebo (sunflower oil as placebo for Omega3 fatty acids; isomaltulosio as placebo for Anthocyanins and Alpha-cyclodextrins)
  Interventions: Behavioral: diet; Other: placebo

INTERVENTIONS:
Dietary Supplement: omega-3 fatty acids, anthocyanins and alpha-cyclodextrins — administration for 12 weeks
  Arms: intervention
Behavioral: diet — 12 weeks of personalized diet according to the Mediterranean standard diet referrals, the Healthy Eating Plate recommendations of Harvard University School of Public Health, and the reference intake levels of nutrients and energy for the Italian population (LARN) for pregnant women
Other: placebo — sunflower oil as placebo for Omega3 fatty acids; isomaltulosio as placebo for Anthocyanins and Alpha-cyclodextrins; administration for 12 weeks
  Arms: placebo

SUMMARY:
Our trial aims to assess the effect of nutraceutical supplements (omega-3 fatty acids, anthocyanins and alpha-cyclodextrins) in patients affected by gestational diabetes.

Pregnant women with gestational diabetes at 24-28 weeks of gestation are enrolled in a double-blind trial and randomized to receive either nutraceutical supplements or a placebo for 12 weeks.

DETAILED DESCRIPTION:
Randomized, Double-blind trial Aims: evaluation of the metabolic effect on patients affected by gestational diabetes of anti-inflammatory, anti-oxidant nutraceutical supplementation with omega-3 fatty acids, anthocyanins and alpha-cyclodextrins for 12 weeks associated with appropriate nutritional coaching versus nutritional coaching and placebo.

All women receive a personalized diet by a nutrition expert educator and should monitor capillary blood glucose levels. Patients receive twice-weekly antenatal testing, including ultrasonography for fetal growth and well-being maternal weight body fat mass distribution evaluation using skinfold caliper, dietary counselling. Blood and urine samples are drawn from all patients at recruitment and at the last study visit.

ELIGIBILITY:
Inclusion Criteria:

* patients between 24 and 28 weeks of gestation with positive result to an Oral Glucose Tolerance Test with 75 gr glucose performed after 24 gestational weeks, according to the International Association of Diabetes and Pregnancy Study Group (IADPSG) recommendations (at least one of the following criteria: baseline glycemia ≥ 92 mg/dl, 1-h glycemia ≥ 180 mg/dl, 2-h glycemia ≥ 153 mg/dl)
* maternal age ≥ 18 years.

Exclusion Criteria:

* multiple pregnancies
* fetal malformation
* maternal diseases (type 1 and type 2 diabetes, hypothyroidism and hyperthyroidism, immunological disorders)
* abnormal blood glucose values before 24 weeks of gestation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant patients
Enrollment: 51 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
capillary blood glucose level | 12 weeks
  percentage of patients with median capillary blood glucose values 10 mg/dl below the target (if the fetal abdominal circunference is below 75° percentile according to gestational age: basal level 95 mg/dl, 2-h post prandial level 120 mg/dl; if the fetal abdominal circunference is above 75° percentile according to gestational age: basal level 90 mg/dl, 2-h post prandial level 110 mg/dl;
plasmatic glycated haemoglobin | 12 weeks
  change in plasmatic glycated haemoglobin

SECONDARY OUTCOMES:
therapy for diabetes | 12 weeks
  percentage of patients requiring pharmacological treatment for gestational diabetes such as insulin or methformin

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Ferrazzi, Professor, Study Director — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: No